CLINICAL TRIAL: NCT05789732
Title: Efficacy of Silodosin, Tadalafil Alone Versus Silodosin Plus Tadalafil as Medical Expulsive Therapy for Lower Ureteric Stones: A Prospective Randomized Placebo Controlled Study
Brief Title: Silodosin, Tadalafil Alone vs. Silodosin Plus Tadalafil as MET for Lower Ureteric Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tamer Abd El-Wahab Diab, Lecturer of Urology, Faculty of Medicine, Benha University, Benha, Egypt, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rc 22-3-2023
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Lower Ureteric Stones; Medical Expulsive Therapy; Tadalafil; Silodosin
MeSH Terms: interventions — silodosin; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo group (Placebo Comparator): Patients in this group will receive placebo treatment once daily.
  Interventions: Drug: Placebo
- Silodosin group (Experimental): Patients will receive Silodosin 8 mg once daily.
  Interventions: Drug: Silodosin
- Tadalafil group (Experimental): Patients will receive Tadalafil 5 mg once daily.
  Interventions: Drug: Tadalafil
- Silodosin and Tadalafil (Experimental): Patients will receive Silodosin 8mg in combination with Tadalafil 5 mg once daily.
  Interventions: Drug: Silodosin and Tadalafil

INTERVENTIONS:
Drug: Placebo — Patients will receive placebo treatment once daily.
  Arms: Placebo group
Drug: Silodosin — Patients will receive Silodosin 8 mg once daily.
  Arms: Silodosin group
Drug: Tadalafil — Patients will receive Tadalafil 5 mg once daily.
  Arms: Tadalafil group
Drug: Silodosin and Tadalafil — Patients will receive Silodosin 8mg in combination with Tadalafil 5 mg once daily.
  Arms: Silodosin and Tadalafil

SUMMARY:
This study will compare the efficacy of silodosin, tadalafil versus silodosin plus tadalafil as Medical Expulsive Therapy (MET) for lower ureteric stones.

DETAILED DESCRIPTION:
The global incidence of urolithiasis, a disease with a high recurrence rate, is increasing. Urolithiasis is one of the most common disorders of the urinary tract with a lifetime prevalence of up to 15% with men affected three times more than women.

Urolithiasis causes recurrent stone formers to experience a decline in quality of life, and there is an increasing socioeconomic burden associated with the management of urolithiasis. Improved quality of life may also have increased its prevalence. A significant proportion, about 1/5th of urinary tract stones, is found in the ureter, of which 2/3rd is seen in the distal ureter. Initially, a colicky pain of various grades presents with ureteric stone. It is one of the most common problems that compel a patient to an emergency room.

Methods to manage ureteral stones include conservative treatment, pharmacological treatment (e.g., medical expulsive therapy), shock wave lithotripsy, and surgical treatment. Thus, urologists must select the appropriate treatment for each patient (i.e., non-surgical or surgical). Today, medical expulsive therapy has become the most used modality of treatment for urolithiasis. During this treatment, the ureter smooth muscle is treated via various drugs by different mechanisms.

Blocking alpha-(α-) 1 adrenergic receptor, especially in the distal third decreases basal smooth muscle contraction and causes propulsive antegrade peristalsis helping stone expulsion. By increasing the intraureteral pressure gradient around the stone, alpha-1 adrenergic receptor antagonists eject distal ureteral stones.

Significant pathological changes can occur when ureteric stones are impacted. +is can cause an inflammatory reaction with mucosal edema which could further worsen the ureteric obstruction, increasing the risk of impaction and retention. However, selective alpha-1 blockers, such as tamsulosin and silodosin, have been the treatment of choice, with proven efficacy in multiple clinical trials. Silodosin is a more selective α-1A adrenoceptor blocker with a better stone expulsion rate than tamsulosin.

Recently, a newer Phosphodiesterase type 5 inhibitor, tadalafil, has shown action on the nitric oxide-cyclic guanosine monophosphate signaling pathway of smooth muscles, resulting in increased levels of cyclic guanosine monophosphate, causing ureteric relaxation.

Due to its smooth muscle relaxation mechanism, tadalafil has received US Food and Drug Administration approval to treat many urinary tract diseases. Therefore, the combination of silodosin and tadalafil drugs is aimed to facilitate stone passage by better ureteric relaxation and reducing intramural ureter pressure. Although there have been few similar studies using various combinations, comparing the efficacy of silodosin and tadalafil vs. silodosin are very few, and these studies have taken longer duration of treatment (4 to 6 weeks) which might have affected the outcome.

ELIGIBILITY:
Inclusion Criteria:

* 168 patients aged >18 years old.
* Both sexes.
* Diagnosed with lower ureteric stone from 5mm to 10mm in size.

Exclusion Criteria:

* Patients with multiple or bilateral ureteric stones
* single kidney or impairment of renal function
* Urinary tract infection (UTI)
* Marked hydronephrosis
* Patients presenting with severe intractable pain and requiring emergency intervention
* Any urologic anomalies or history of ureteral surgery
* Pregnancy
* Pediatric populations
* Ischemic heart disease
* Congestive cardiac failure
* Complicated hypertension
* Patients on concomitant treatment with nitrates or calcium channel blockers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Stone expulsion rate | Intraoperatively
  Stone expulsion rate will be recorded

SECONDARY OUTCOMES:
Stone expulsion time | Intraoperatively
  Stone expulsion time will be recorded
Amount of analgesia used | Intraoperatively
  The amount of analgesia used will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospitals, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study will be available under a reasonable request of the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the end of the study